THE EFFECT OF HFNC ON MORTALITY AND ICU STAY TIME IN ACUTE RESPIRATORY FAILURE DUE TO COVID-19 PNEUMONIA

06.06.2020

## **Statistical Analysis:**

The data were evaluated using the Windows SPSS 22 package program. Descriptive findings number and percentage distributions for categorical variables; numerical variables are given as mean and standard deviation.

As statistical analysis, Mann-Whitney U test was used for categorical variables, chi-square, normal distribution conditions for numerical variables, Kolmogorov-Simirnov, histogram, and Q-Q Plots graph. Significance level was accepted as p <0.05.